CLINICAL TRIAL: NCT00684814
Title: A Randomized, Two-way Crossover, Single-Dose, Open-Label Study to Evaluate the Relative Bioequivalence of a Test Tablet Formulation of Zolpidem Tartrate 10 mg, Compared to an Equivalent Dose of Ambien® in Healthy Adult Subjects.
Brief Title: Bioequivalence Study of Zolpidem Tartrate Tablets and Ambien® Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President R&D, Mutual Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 04064
Record Dates: First submitted 2008-05-24; First posted 2008-05-28 (Estimated); Results first posted 2010-01-08 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: equivalency; Therapeutic equivalency
MeSH Terms: interventions — Zolpidem; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zolpidem Tartrate 10 mg Tablets (Experimental): A single dose of zolpidem tartrate 10 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Zolpidem Tartrate 10 mg tablet
- Zolpidem Tartrate (Ambien®) 10 mg Tablets (Experimental): A single dose of Ambien® 10 mg administered after an overnight fast of at least 10 hours.
  Interventions: Drug: Zolpidem Tartrate 10 mg tablet (Ambien®)

INTERVENTIONS:
Drug: Zolpidem Tartrate 10 mg tablet — 10 mg tablet administered after an overnight fast of at least 10 hours
  Arms: Zolpidem Tartrate 10 mg Tablets
Drug: Zolpidem Tartrate 10 mg tablet (Ambien®) — 10 mg tablet administered after an overnight fast of at least 10 hours
  Other Names: Ambien®, Sanofi-Synthelabo Inc.
  Arms: Zolpidem Tartrate (Ambien®) 10 mg Tablets

SUMMARY:
The purpose of this study is to compare the bioequivalence of a test formulation of zolpidem tartrate tablets to an equivalent oral dose of the commercially available reference drug product Ambien® (zolpidem tartrate tablets) in adult subjects under fasted conditions.

DETAILED DESCRIPTION:
The purpose of this study is to compare the bioequivalence of a test formulation of zolpidem tartrate tablets to an equivalent oral dose of the commercially available reference drug product Ambien® (zolpidem tartrate tablets) in adult subjects under fasted conditions.

Thirty-eight healthy, non-smoking, non-obese male and female volunteers at least 18 years of age will be randomly assigned in a crossover fashion to receive each of two zolpidem tartrate dosing regimens in sequence with a 7 day washout period between dosing periods. On the morning of Day 1, after an overnight fast of at least 10 hours, subjects will receive either a single oral dose of the test formulation, zolpidem tartrate (1 x 10 mg tablet) or a single oral dose of the reference formulation, Ambien® (1 x 10 mg tablet). After a 7 day washout period, on the morning of Day 8 after an overnight fast, subjects will receive the alternate regimen. Blood samples will be drawn from all participants before dosing and for 12 hours post dose at times sufficient to adequately define the pharmacokinetics of zolpidem tartrate. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout the confinement portion of the study for adverse reactions to the study drugs and/or procedures. Blood pressure and pulse rate will be obtained prior to dosing and at 0.5, 1, 2, 4 and 12 hours post-dose. All adverse events whether elicited by query, spontaneously reported or observed by clinic staff will be evaluated by the investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male or Female; similar proportions of each preferred
* Age: At least 18 years
* Weight: must be 15% of ideal weight for height and frame
* Subjects must be in good health and physical condition as determined by medical history
* Subjects must read and sign the Consent Form

Exclusion Criteria:

* History of treatment for alcoholism, substance abuse, or drug abuse within past 24 months.
* History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
* History of GERD, malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
* History of treatment for asthma within the past five (5) years.
* History of mental depression.
* History of pulmonary disease.
* History of sleep apnea.
* Females who are pregnant or lactating.
* History of hypersensitivity to zolpidem tartrate, or any hypnotic or sedative.
* Treatment with any other investigational drug during the four weeks prior to the initial dosing of the study.
* Donation of blood within four weeks prior to the initial dosing of the study
* Smokers or subjects who use tobacco/nicotine products. Three months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2004-05; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

REFERENCES:
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets: On the morning of Day 1 after an overnight fast of at least 10 hours, each subject received one tablet of the test formulation, zolpidem tartrate 10 mg, followed by a 7 day washout period. Then, on the morning of Day 8 after an overnight fast of at least 10 hours, each subject received a single tablet of the reference formulation, Ambien® 10 mg.
- Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets: On the morning of Day 1 after an overnight fast of at least 10 hours, each subject received one tablet of the reference formulation, Ambien® 10 mg, followed by a 7 day washout period. Then, on the morning of Day 8 after an overnight fast of at least 10 hours, each subject received a single tablet of the test formulation, zolpidem tartrate 10 mg.
Period: First Intervention
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Washout Period of 7 Days
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 19 | 19
Completed | 17 | 15
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Intervention
Arm/Group | Zolpidem Tartrate 10 mg Tablets Then Ambien® 10 mg Tablets | Ambien® 10 mg Tablets Then Zolpidem Tartrate 10 mg Tablets
Started | 17 | 15
Completed | 16 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zolpidem Tartrate 10 mg Tablets and Ambien® 10 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either zolpidem tartrate 10 mg or Ambien® 10 mg following an overnight fast of at least 10 hours.
Arm/Group | Zolpidem Tartrate 10 mg Tablets and Ambien® 10 mg Tablets
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.92 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) for Zolpidem Tartrate
Description: The maximum or peak concentration that zolpidem tartrate reaches in the plasma.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing (hour 0), and then at 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 4, 5, 6, 8, 10, and 12 hours after dose administration
Population: Plasma concentration data for 31 of 38 participants were used in the statistical analysis. Six subjects dropped from study period I and one subject dropped from study period II.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Zolpidem Tartrate 10 mg Tablets: Each subject received one tablet of zolpidem tartrate 10 mg after an overnight fast of at least 10 hours.
- Ambien® 10 mg Tablets: Each subject received one tablet of Ambien® 10 mg after an overnight fast of at least 10 hours.
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 31 | 31
ng/mL | 191.94 (74.77) | 193.43 (59.95)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)] for Zolpidem Tartrate
Description: The area under the plasma concentration versus time curve, from time 0 to the time of the last measurable zolpidem tartrate concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 31 | 31
ng-hr/mL | 682.17 (285.78) | 692.47 (290.89)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]for Zolpidem Tartrate
Description: The area under the zolpidem tartrate plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable plasma concentration to the elimination rate constant.
Time Frame: serial pharmacokinetic blood samples drawn prior to dosing (hour 0), then 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.25, 2.5, 2.75, 3, 3.25, 3.5, 4, 5, 6, 8, 10, and 12 hours after dose administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng-hr/mL
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Number analyzed (Participants) | 31 | 31
ng-hr/mL | 723.14 (327.83) | 739.63 (351.51)

ADVERSE EVENTS:
Groups:
- Zolpidem Tartrate 10 mg Tablets; Ambien® 10 mg Tablets: All subjects received each of the two study regimens in a randomly assigned sequence of dosing periods. On the mornings of Day 1 and Day 8, each subject received one tablet of either zolpidem tartrate 10 mg or Ambien® 10 mg following an overnight fast.
Arm/Group | Zolpidem Tartrate 10 mg Tablets | Ambien® 10 mg Tablets
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/36
Other Adverse Events (participants affected / at risk) | 10/34 | 14/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zolpidem Tartrate 10 mg Tablets (N=34) | Ambien® 10 mg Tablets (N=36)
Achy joints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 6 (6) | 6 (6)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Unsteadiness (Nervous system disorders) | 3 (3) | 1 (1)
Hiccups (Gastrointestinal disorders) | 3 (3) | 5 (6)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Head cold (Infections and infestations) | 0 (0) | 1 (1)
Tightness in lungs (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Confusion (Nervous system disorders) | 1 (1) | 1 (1)
Slurred speech (Nervous system disorders) | 0 (0) | 1 (1)
Visual disturbances (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days